CLINICAL TRIAL: NCT02783313
Title: Clinical Effectiveness of Standard Versus Pathogen-reduced Buffy Coat-derived Platelet Concentrates in Plasma in Hemato-oncological Patients.
Brief Title: Pathogen Reduction Evaluation & Predictive Analytical Rating Score
Acronym: PREPAReS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sanquin Research & Blood Bank Divisions (Other)
Collaborators: Terumo BCT (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ABR30643; NTR2106 (Registry Identifier: Dutch Trial Register)
Record Dates: First submitted 2016-04-11; First posted 2016-05-26 (Estimated); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Thrombocytopenia
Keywords: pathogen inactivation; platelets
MeSH Terms: conditions — Thrombocytopenia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PR-plasma-PCs (Experimental): Pooled buffy coat-derived pathogen reduced plasma-stored platelet concentrates (PR-plasma-PCs)
  Interventions: Device: Pathogen reduced plasma-stored platelet concentrates
- Plasma-PCs (Active Comparator): Pooled buffy coat-derived plasma-stored platelet concentrates (plasma-PCs)
  Interventions: Other: Plasma-stored platelet concentrates

INTERVENTIONS:
Device: Pathogen reduced plasma-stored platelet concentrates — Platelet concentrates treated with the Mirasol PRT system (pathogen reduction technology) and stored in plasma.
  Arms: PR-plasma-PCs
Other: Plasma-stored platelet concentrates — Platelet concentrates stored in plasma
  Arms: Plasma-PCs

SUMMARY:
The objective of this study is to determine if pooled buffy coat-derived pathogen reduced plasma-stored platelet concentrates are non-inferior compared to plasma-stored platelet concentrates in terms of WHO bleeding complications in hemato-oncological patients with thrombocytopenia.

DETAILED DESCRIPTION:
Currently some pathogen-reduced platelet products (PR-PCs) have passed phase III studies, are in progress or can be expected in the near future. At present some transfusion centers throughout Europe have implemented PR-PCs, but as yet PR-PCs are not formally accepted as a standard product that should be applied nation-wide. Because many uncertainties currently exist on the "optimal" platelet product, it is in the interest of patients, health care providers and the transfusion provider (Sanquin) to decide on evidence.

With all the current safety measures remaining in place, pathogen reduction provides a safety benefit by reducing the number of transfusions of platelet concentrates contaminated with bacteria, but which were missed by the screening method. In the Dutch situation, morbidity is estimated to be 1:14,000 platelet concentrates [Te Boekhorst, Transfusion 2005]. In this publication, two cases of transmission of B. cereus by a platelet transfusion are reported, where both patients experience a life-threatening sepsis, but recover eventually. Cases of bacterial transmission however often go unnoted, so a frequency as low as 1:130,000 has been reported [Dumont, Transfusion 2010]. The same is true for mortality; this value ranges from 1:50,000 to 1:500,000.

A more precautionary benefit is protection against known and unknown pathogens. It is difficult to estimate the actual risk, and consequently to estimate the benefit for the patient. While in The Netherlands no epidemics have occurred against which no screening tests could be developed, including Q-fever, there is a small but real risk that an epidemic can wipe out the blood supply in a country. This has happened in La Réunion, where an epidemic of chikungunya virus urged import of blood products from abroad, followed by rapid introduction of a pathogen reduction technology to ensure the blood supply [Rasongles, Transfusion 2009]. An outbreak of this virus in Italy resulted in suspension of blood collections in an affected area, which led to a low blood inventory as well as a reduced delivery of plasma to fractionation institutes.

Appreciating the difficulties of extrapolating in vitro tests towards in vivo efficacy, platelet products should be tested in clinical trials. Of note, radiolabeling techniques in volunteers as required by the FDA, are not used in the Netherlands. For major product variations in the Netherlands, investigators depend on studies in patients. Extending storage for logistic purposes, combined with maintaining or even improving the safety of platelet products, and maintaining clinical efficacy are the main features in the development of new platelet products. In this study protocol, the aim is to investigate transfusion efficacy of two different platelet products: plasma-PCs, and pathogen-reduced (PR)-plasma-PCs, combining extended storage with or without treatment with a photochemical pathogen reduction technique. Prior to the start of the clinical study an in vitro study of the product has been performed, showing that the study product meets the current in vitro quality requirements for release for transfusion. However, on site implementation validation still has to take place.

Refractoriness to platelet transfusions and bleeding complications are the main clinical problems in intensively treated hemato-oncological patients and are essential endpoints for transfusion studies as well. In this trial, bleeding will be scored according to the World Health Organization (WHO) scale as a primary endpoint. Refractoriness is defined as a 1-hour CCI <7.5 and/or a 24-hour CCI <4.5 after ABO compatible platelet transfusions on at least two successive occasions. Known causes of non-alloimmune refractoriness are included in this trial because for the purpose of generalization, relevant to develop a national product, testing transfusion efficacy of new platelet products should imply all patients in need of a preventive support with platelet transfusions. The 1- and 24-hour CCI are commonly used to evaluate platelet transfusions and, albeit not without discussion, currently the platelet count is the only parameter in trigger-based transfusion policy. The ratio of both the 1-hour and 24-hour CCI mirrors both platelet recovery immediately after transfusion as the 1-hour CCI, and platelet survival one day after transfusion as the 24-hour CCI. Other secondary clinical endpoints of the trial will be transfusion requirement (red cells and platelets), transfusion interval to next transfusion and adverse reactions.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. Expected ≥ 2 platelet transfusion requirements;
3. Signed informed consent;
4. Having hemato oncological disease including those who undergo myelo ablative allogeneic stem cell transplant therapy.

Exclusion Criteria:

1. Micro-angiopathic thrombocytopenia (TTP, HUS) and ITP;
2. Bleeding > grade 2 at randomization ( after treatment, the patient can be randomized in the study after 2 or more weeks after the last transfusion that was used to stop the bleeding);
3. Known immunological refractoriness to platelet transfusions;
4. HLA- and/or HPA-allo immunization and/or clinical relevant auto-antibodies;
5. Indications to use hyper-concentrated (plasma-reduced) platelet concentrates, i.e. patients with known severe allergic reactions and documented transfusion-associated circulatory overload (TACO);
6. Pregnancy (or lactating);
7. Prior treatment with pathogen-reduced blood products;
8. Known allergy to riboflavin or its photoactive products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 567 (Actual)
Dates: Start 2010-11-17; Primary Completion 2016-04-30 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with WHO grade ≥ 2 bleeding complications | Transfusion episode (from the day of the first on-study transfusion until study completion), an average of 20 days
  Any WHO grade ≥ 2 bleeding event, as determined by daily assessment of bleeding symptoms, and documentation of any red blood cell transfusions to treat bleeding

SECONDARY OUTCOMES:
1 and 24 hour count increment | 1 and 24 hours post-transfusion
1 and 24 hour corrected count increment (CCI) | 1 and 24 hours post-transfusion
(1+24 hour CCI)/2 | 1 and 24 hours post-transfusion
Adverse transfusion reactions | On-study episode (from the day of randomization until study completion), an average of 25 days
  All transfusion-associated side effects observed within 6 hours after platelet transfusion
Total transfusion requirement of red cells and platelets | Transfusion episode (from the day of the first on-study transfusion until study completion), an average of 20 days
  Number of occurrences of a platelet transfusion or a red cell transfusion among subjects who have had at least one platelet transfusion
Platelet transfusion interval | Transfusion episode (from the day of the first on-study transfusion until study completion), an average of 20 days
  Time in hours between the last and first occurrence of a platelet transfusion, divided by the number of platelet transfusion occurrences minus 1, among subjects who have had at least two platelet transfusions
Rate of HLA allo-immunization | From the day of randomization until 56 days after randomization
In vitro quality markers related with the 1-hour or 24-hour CCI | 1 and 24 hours post-transfusion
Clinical factors interacting on primary endpoint, including in vivo variables of immunological responses; and of hemostasis in the recipients after transfusion as compared prior to transfusion. | Transfusion episode (from the day of the first on-study transfusion until study completion), an average of 20 days
  Severity of the WHO bleeding grade as determined by daily assessment of bleeding symptoms, related to the level of circulating HLA allo antibodies as determined in a blood sample collected every week during the on-study episode; severity of the WHO bleeding grade as determined by daily assessment of bleeding symptoms at the day of occurrence of a platelet transfusion as compared to the day after the occurrence of a platelet transfusion

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis Kerkhoffs, MD, PhD, Principal Investigator — Sanquin Blood Bank
Locations (10):
- Canada (5):
  - McMaster University, Hamilton
  - Kingston General Hospital, Kingston
  - London Health Sciences Centre, London
  - Ottawa Hospital, Ottawa
  - Sunnybrook Health Sciences Centre, Toronto
- Netherlands (4):
  - Leiden University Medical Center, Leiden
  - Maastricht University Medical Center, Maastricht
  - Erasmus Medical Center, Rotterdam
  - Haga Ziekenhuis, The Hague
- Haukeland University Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ypma PF, van der Meer PF, Heddle NM, van Hilten JA, Stijnen T, Middelburg RA, Hervig T, van der Bom JG, Brand A, Kerkhoffs JL; PREPAReS Study Group. A study protocol for a randomised controlled trial evaluating clinical effects of platelet transfusion products: the Pathogen Reduction Evaluation and Predictive Analytical Rating Score (PREPAReS) trial. BMJ Open. 2016 Jan 27;6(1):e010156. doi: 10.1136/bmjopen-2015-010156. PMID 26817642
- [Result] van der Meer PF, Ypma PF, van Geloven N, van Hilten JA, van Wordragen-Vlaswinkel RJ, Eissen O, Zwaginga JJ, Trus M, Beckers EAM, Te Boekhorst P, Tinmouth A, Lin Y, Hsia C, Lee D, Norris PJ, Goodrich RP, Brand A, Hervig T, Heddle NM, van der Bom JG, Kerkhoffs JH. Hemostatic efficacy of pathogen-inactivated vs untreated platelets: a randomized controlled trial. Blood. 2018 Jul 12;132(2):223-231. doi: 10.1182/blood-2018-02-831289. Epub 2018 May 17. PMID 29773572